CLINICAL TRIAL: NCT05836545
Title: A Randomized, Single-Blind, Investigator Initiative Trial Study of Remimazolam Versus Midazolam for Sedation in Diagnostic Upper Gastrointestinal Endoscopy
Brief Title: Remimazolam Versus Midaszolam for Sedation in Diagnostic Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-08-2391
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam (Active Comparator): The patient with midazolam
  Interventions: Drug: Midazolam
- Remimazolam (Experimental): The patient with remimazolam
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — The patient with remimazolam
  Arms: Remimazolam
Drug: Midazolam — The patient with midazolam
  Arms: Midazolam

SUMMARY:
The goal of this clinical trial is to compare the efficacy of remimazolam with midazolam in patients undergoing gastrointestinal endoscopy. The main questions it aims to answer are:

* Superiority of total procedure time in remimazolam compared to midazolam
* The success of sedation time

This is the single blind study.; Patients will not know what they are given as the sedation drug If there is a comparison group: Researchers will compare patients with midazolam group to see if remimazolam group is superior to midazolam group

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed for this clinical trials
* Patients who want diagnostic endoscopy under sedation
* The total procedure time which is predicted within 15 minutes
* ASA >=2
* BMI more than 18.5kg/m2, less than 30kg/m2

Exclusion Criteria:

* Patients who have stomach illness
* Patients with respiratory disease
* Mallampati Score>=3
* Systolic BP >160mmHg or <90mmHg
* Refractory Hypertension
* Uncontrolled glaucoma
* Severe liver failure or chronic kidney disease
* Patients with drug abuse or alcohol abuse within 1 year
* Patients who are sensitive for certain medication (such as benzodiazepine, remimazolam)
* Obstructive sleep dyspnea patients
* Galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Pregnant, breast feeding patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Total procedure time | begin when the drug is give to when the endoscopy is withdrawn

SECONDARY OUTCOMES:
The success rate of sedation | Completion of the whole endoscopy procedures, No requirement for an alternative and/or rescue sedative, Administered up to a maximum of five supplemental doses within 15 mnutes after the initial dose

CONTACTS AND LOCATIONS:
Overall Officials: Taejun Kim, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park Y, Lee JK, Lee KH, Kim T, Kang SH, Ahn DW, Kim SB, Kim SJ. Remimazolam Enables Faster Sedation Induction and Recovery Compared With Midazolam in Diagnostic Upper Gastrointestinal Endoscopy: A Multicenter Randomized Controlled Trial. United European Gastroenterol J. 2026 Feb;14(1):e70147. doi: 10.1002/ueg2.70147. Epub 2025 Nov 24. PMID 41284133